CLINICAL TRIAL: NCT04905849
Title: Enhancing Cognitive Control Abilities Using Mobile Technology in a Senior Living Community
Acronym: ACCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic prevented the participating senior centers from recruiting as originally stipulated
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AG058896 (NIH); R21AG058896 (NIH)
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Aging; Cognitive Change

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive Cognitive Control Trainer (ACCT) (Experimental): There are three modules within the game, each training a different aspect of cognitive control (attention, goal management, working memory): a visual search task for attention abilities, a spatial span task for working memory, and a task switching paradigm for goal management abilities. There are also 3 different levels of difficulty associated with each module; advancing to the next level delivers an advanced challenge that enhances the difficulty in performing the given cognitive task. Participants advance to the next level of difficulty following 6 training sessions occurring over 2 weeks, with the total training experience being 6 weeks of training (3 days/week), with each training session lasting 36 minutes (not including self-paced breaks).
  Interventions: Behavioral: Adaptive Cognitive Control Trainer (ACCT)
- Active Control Group (Active Comparator): An active control application will be used for this arm. The total training experience here will also be for 6 weeks (3 days/week), with each training session lasting ~30 minutes (not including self-paced breaks). Here an app that is matched in terms of expectancy of benefits compared to our training groups will be determined by questioning 100 naïve individuals to predict their expected improvement on each cognitive domain across a multitude of possible applications.
  Interventions: Behavioral: Active Control App

INTERVENTIONS:
Behavioral: Adaptive Cognitive Control Trainer (ACCT) — Module 1: Attention=> This module demands an active scan of the screen in search for a target, much like traditional visual search tasks. Participants quickly identify the direction that a probe target is facing (up, down, left, right), and are aided by the presence of directional cue indicating where the location of the target will appear.
  Module 2: Goal Management=> Requires participants to rapidly switch their focus based on distinct rules. Participants are presented with exemplar objects along with a target, and are asked to indicate which exemplar presented is most like the target.
  Module 3: Working Memory=> Engages spatial working memory resources similar to the Corsi block task. Participants memorize the location of objects on screen followed by a 5-7 second delay period, with a correct response leading to a greater number of potential targets to be memorized on the next trial (and vice versa).
  Arms: Adaptive Cognitive Control Trainer (ACCT)
Behavioral: Active Control App — The app used here is undergoing expectancy-matching at the present time, will be updated with the final app characteristics when completed out of a list of several possibilities
  Arms: Active Control Group

SUMMARY:
The goal of this study is to test the feasibility of launching a personalized digital health assessment and remediation program for the older adults in senior living communities based upon an initial characterization of these abilities. Evidence of feasibility here using these unique methodological approaches would provide empirical evidence supporting the basis for a larger-scale implementation of such digital health technologies into less controlled senior settings.

ELIGIBILITY:
Inclusion Criteria:

* Must be living at a Senior Living Community
* have own iPad and/or smartphone,
* native-English speaker.

Participation across a spectrum of cognitive abilities is desired for this study, specifically for older adults in a community setting.

Exclusion Criteria:

* Do not have any physical or cognitive limitations that would clearly prevent them from utilizing these applications as intended

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Anguera, Ph.D., Principal Investigator — UC San Francisco
Locations (1):
- UC San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adaptive Cognitive Control Trainer (ACCT) | Active Control Group
Started | 12 | 0
Completed | 6 | 0
Not Completed | 6 | 0
Not completed — The COVID pandemic devastated this study, as Brookdale efforts focused on resident health and safety | 6 | 0

BASELINE CHARACTERISTICS:
Population: Participants from different Brookdale Senior Living Communities across the United States
Groups:
- Total: Total of all reporting groups
Arm/Group | Adaptive Cognitive Control Trainer (ACCT) | Active Control Group | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (5.5) |  | 72 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 4 |  | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ACE-X [Count of Participants; unit: Participants] — ACE-X is an iOS app measuring cognitive control, specifically attention and working memory abilities including a version of a Continuous Performance Task (CPT) and a foward/backward spatial span task (Corsi Block). For the CPT like task, the measure of interest per participant was mean accuracy (% of trials that were correctly responded to) and response time variability (the variance associated with response time). For the Span tasks, the measure of interest was the maximum length of the span achieved. Here our goal was to measure HOW MANY participants were able to complete the ACE-X tasks.
  Participants
    CPT- | 6 | 0 | 6
    Spatial Span | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Attempted to Complete the Adaptive Cognitive Evaluation (ACE) From Baseline at 6 Weeks
Description: ACE is a custom mobile cognitive health assessment battery that presents paradigms typically used in standard cognitive neuroscience laboratories. Here the investigators will assess a measure of (1) Attention and (2) Working memory in the ACE software.
Time Frame: At Baseline and post intervention at the 6 week mark
Population: Individuals from Brookdale Senior Living Communities from across U.S. We counted How Many participants attempted to complete the ACE-X battery.
Measure: Count of Participants; unit: Participants
Arm/Group | Adaptive Cognitive Control Trainer (ACCT) | Active Control Group
Number analyzed (Participants) | 6 | 0
Participants | 6 | 0

2. Secondary Outcome: Mean Performance on the Everyday Cognition Scale (ECog) From Baseline at 6 Weeks
Description: The Everyday Cognition Scale (ECog) measures the ability to perform everyday tasks that demand memory, language, visuospatial abilities, planning, organization, and divided attention. The ECog consists of a global and domain scores for each of the previously described categories, and is scored as follows: 1= better or no change compared to 10 years earlier, 2= questionable/occasionally worse compared to 10 years earlier, 3= consistently a little worse compared to 10 years earlier, 4= consistently much worse compared to 10 years earlier. Thus, the lower the overall score is on this measure at both the global and domain score level, the better one is performing with respect to their cognition.
Time Frame: At Baseline and post intervention at the 6 week mark
Population: This measure was not collected in the end; none of the participants completed this measurement
Units Other Than Participants: survey count
Groups:
- Adaptive Cognitive Control Trainer (ACCT): There are three modules within the game, each training a different aspect of cognitive control (attention, goal management, working memory): a visual search task for attention abilities, a spatial span task for working memory, and a task switching paradigm for goal management abilities.
  Adaptive Cognitive Control Trainer (ACCT): Module 1: Attention=> This module demands an active scan of the screen in search for a target, much like traditional visual search tasks. Participants quickly identify the direction that a probe target is facing (up, down, left, right), and are aided by the presence of directional cue indicating where the location of the target will appear.
  Module 2: Goal Management=> Requires participants to rapidly switch their focus based on distinct rules. Participants are presented with exemplar objects along with a target, and are asked to indicate which exemplar presented is most like the target.
  Module 3: Working Memory=> Engages spatial working memory resources similar to the Corsi block task. Participants memorize the location of objects on screen followed by a 5-7 second delay period, with a correct response leading to a greater number of potential targets to be memorized on the next trial (and vice versa).
Arm/Group | Adaptive Cognitive Control Trainer (ACCT) | Active Control Group
Number analyzed (Participants) | 0 | 0
Number analyzed (survey count) | 0 | 0

3. Secondary Outcome: Mean Change on Cognitive Failures Questionnaire (CFQ) From Baseline at 6 Weeks
Description: The Cognitive Failures Questionnaire (CFQ) assesses participant distractibility. The CFQ score ranges from 0 to 100, with the lower the overall score is on this measure, the better one is performing with respect to their cognition.
Time Frame: At Baseline and post intervention at the 6 week mark
Population: No data was collected in the end for this measure, as no participants completed this measure.
Arm/Group | Adaptive Cognitive Control Trainer (ACCT) | Active Control Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change on General Health and Well-being (SF-36) From Baseline at 6 Weeks
Description: The general health and well-being (SF-36) score assesses participant health. The SF-36 score ranges from 0 to 100. The higher the overall score is on this measure, the better one is performing with respect to their health and well-being.
Time Frame: At Baseline and post intervention at the 6 week mark
Population: Note that no data was collected for this measure, as none of the participants completed this requested survey.
Arm/Group | Adaptive Cognitive Control Trainer (ACCT) | Active Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The time frame was over the course of the study (e.g. 1 year) Note that the study took place over a 6 week period, with 1 week given as a window to complete each assessment period Baseline -> 4 week intervention -> Post-training Assessment This was the time period over which adverse event data were collected
Description: We used the same definition used by clinicaltrials.gov. Participants were asked to self-report any adverse events over the course of the study.
Arm/Group | Adaptive Cognitive Control Trainer (ACCT) | Active Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12 | 0/0

LIMITATIONS AND CAVEATS:
The primary limitation was the onset of COVID pandemic, which prevented the study from being completed entirely, in any way, like the originally designed study. This restricted the amount, quality, and extent of data collected. Our partners at Brookdale acknowledged that they would not be able to contribute to this project as desired as "we're trying to keep our seniors alive right now, and do not have the bandwidth to help with any other endeavors"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04905849/Prot_SAP_000.pdf